CLINICAL TRIAL: NCT06977360
Title: Feasibility, Acceptability and Preliminary Efficacy of the New Iteration of the Innovative Smartphone-based Care Solution for Women With Breast Cancer Undergoing Chemotherapy (iCareBreast+): A Pilot Study Research Proposal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Buddy Healthcare Ltd OY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: iCareBreast+
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Digital Health; mHealth; Mobile health; Psychosocial; Randomized Controlled Trial; Self-efficacy; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental)
  Interventions: Other: Routine care
- Intervention Group (Experimental)
  Interventions: Other: Routine care + iCareBreast+ mobile app

INTERVENTIONS:
Other: Routine care — Routine care provided by NCCS
  Arms: Control Group
Other: Routine care + iCareBreast+ mobile app — Routine care provided by NCCS (identical to the control group) along with access to the iCareBreast+ mobile app
  Arms: Intervention Group

SUMMARY:
The overall aim of the study is to evaluate the feasibility, acceptability and preliminary effects of the next iteration of iCareBreast+, an innovative breast care e-support intervention programme, by refining existing contents and building new contents based on comprehensive assessment of breast cancer women's needs and preferences among breast cancer patients undergoing chemotherapy.

The specific objectives of this study are:

1. To develop a new iteration of an innovative smartphone-based self-care solution for patients with breast cancer undergoing chemotherapy (iCareBreast+);
2. To assess the feasibility and acceptability of iCareBreast+; and
3. To explore the preliminary effects of iCareBreast+ on the primary outcome of self-efficacy, and knowledge of breast cancer treatment, as well as secondary outcomes including anxiety, depression, health-related quality of life (HRQoL), social support and satisfaction with oncologic care.

DETAILED DESCRIPTION:
A two-group pilot randomized controlled trial with pretest and post-test will be conducted in a tertiary hospital in Singapore. Women with breast cancer requiring chemotherapy (n = 40) will be recruited and randomly allocated to the intervention group (receiving iCareBreast+ and routine care) or the control group (routine care only). Feasibility data (patient recruitment and attrition, usefulness, ease of use, strengths and weaknesses), as well as app quality data will be collected. Health outcomes will be measured using validated instruments at baseline and immediately after the 2-month intervention.

ELIGIBILITY:
Inclusion Criteria:

Women who:

* are the age of 21 years old and above at the point of recruitment;
* are diagnosed with stage 1-3 breast cancer;
* will undergo chemotherapy first time (initiating or up to #4 cycles of chemo is acceptable);
* can speak, read and write in English or Mandarin; and
* has access to and able to use smart phone.

Exclusion Criteria:

Those who :

* are with a history of or concurrent other cancer types;
* have been suffering from psychiatric illness (e.g., schizophrenia), anxiety disorder or other mood disorder or impaired cognitive function;
* have alcohol or substance abuse within the previous year;
* are undergoing concurrent psychosocial interventions; and
* have been in the bereavement period in the last 6 months
* are in their pregnancy.

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The feasibility of research method and Intervention | Throughout data collection period, estimated up to six months or until last subject with last visit completion whichever is later.
  Participants recruitment and attrition rates.
The acceptability of intervention | After intervention (two months immediately post intervention)
  Process evaluation (semi-structured interview) and app quality (mobile app rating scale score)
The impact of psychosocial intervention (iCareBreast+ app) on cancer self-efficacy | Baseline (on enrolment day), and after Intervention (two months immediately post intervention)
  Changes of Self-efficacy Score (Self-efficacy Score from the cancer Behaviour Inventory-Brief (CBI-B) survey).
The impact of psychosocial Intervention (iCareBreast+ app) on knowledge of breast cancer treatment | Baseline (on enrolment day), and after Intervention (two months immediately post intervention)
  Changes of knowledge Score (Knowledge Score from a scale of 0-10)

SECONDARY OUTCOMES:
The impact of psychosocial Intervention (iCareBreast+ app) on anxiety and depression | Baseline (on enrolment day), and after Intervention (two months immediately post intervention)
  Changes of anxiety and depression Score (Hospital Anxiety and Depression scale).
The impact of psychosocial Intervention (iCareBreast+ app) on cancer related quality of life | Baseline (on enrolment day), and after Intervention (two months immediately post intervention)
  Changes of Cancer related quality of lief Score (Functional Assessment of Cancer Therapy-Breast (FACT-B))
The impact of psychosocial Intervention (iCareBreast+ app) on cancer self-efficacy | Baseline (on enrolment day), and after Intervention (two months immediately post intervention)
  Changes of Social support Score (The Medical Outcomes Study Social Support Survey).
The impact of psychosocial Intervention (iCareBreast+ app) on satisfaction of oncological care | After Intervention (two months immediately post intervention)
  Satisfaction Score (Satisfaction Score from a single item 6-point Ordinal Descriptive Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ryan Shea YC Tan, MBBS, MRCP(UK), MMed, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes